CLINICAL TRIAL: NCT02003859
Title: Predictive Value of pCLE Findings in Pediatric IBD
Status: Completed | Type: Observational
Sponsor: Scientific Center of Children's Health RAMS (Other)
Collaborators: University of Alberta (Other); Harvard Medical School (HMS and HSDM) (Other)
Responsible Party: Principal Investigator, Anton A. Shavrov, M.D., Scientific Center of Children's Health RAMS
Other Study IDs: SCCH-001
Record Dates: First submitted 2013-11-30; First posted 2013-12-06 (Estimated); Last update posted 2014-11-19 (Estimated); Status verified 2014-11

CONDITIONS: Inflammatory Bowel Disease
Keywords: IBD; Pediatrics; pCLE
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — Optical biopsy
Oversight: Data Monitoring Committee: No

SUMMARY:
Studies over the past two decades have convincingly demonstrated the role of barrier dysfunction in the pathogenesis of inflammatory bowel disease. It previously shown that optical biopsy with probe-based confocal laser endomicroscopy (pCLE) could be used to assess mucosal barrier function. Furthermore, mucosal barrier dysfunction on pCLE was shown to be predictive of disease relapse in adult IBD patients. The purpose of the current study is to determine the predictive value of pCLE findings in pediatric IBD patients.

ELIGIBILITY:
Inclusion Criteria:

* signed informed consent
* patients with established IBD

Exclusion Criteria:

* Any kind of allergy
* Bronchial asthma
* Liver or kidney disease
* Inability to sign informed consent

Ages: 10 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric patients with IBD from all over Russia, treated from IBD in our Center
Sampling Method: Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2010-11; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Primary study end-point was moderate to severe flare requiring hospitalization after pCLE | follow up period was a median of 18 months (range 4 to 33)
  The purpose of the current study is to determine the predictive value of pCLE findings in pediatric IBD patients.

CONTACTS AND LOCATIONS:
Overall Officials: Andrey A Shavrov, M.D., Study Chair — The Scientififc Center of Children's Health
Locations (1):
- The Scientific Center of Children's Health, Moscow, Russia

REFERENCES:
- [Derived] Shavrov A, Kharitonova AY, Davis EM, Claggett B, Morozov DA, Brown DK, Shavrov AA, Liu JJ. A Pilot Study of Confocal Laser Endomicroscopy to Predict Barrier Dysfunction and Relapse in Pediatric Inflammatory Bowel Disease. J Pediatr Gastroenterol Nutr. 2016 Jun;62(6):873-8. doi: 10.1097/MPG.0000000000001022. PMID 26513619